CLINICAL TRIAL: NCT06745310
Title: Comparison of Activities of Daily Living and Upper Extremity Exercise Capacity of Individuals with High Body Mass Index with Those with Normal Body Mass Index
Brief Title: Activities of Daily Living and Upper Extremity Exercise Capacity of Individuals with High Body Mass Index
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-20/174
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Body Mass Index; Body Mass Index 25 or Greater; Body Mass Index, Normal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals with high body mass index
- Individuals with normal body mass index

SUMMARY:
Individuals with high and normal body mass index will be included in this study.

ELIGIBILITY:
Inclusion Criteria for individuals with high body mass index:

* Body mass index ≥ 25 kg/m2
* Volunteering for the study

Exclusion Criteria for individuals with high body mass index:

* Having uncontrolled hypertension, diabetes mellitus
* Having comorbidities that may affect physical functions
* Failure to cooperate with tests to be performed
* Liver disease, kidney disease, cancer, lung diseases and serious cardiomyopathies, neurological diseases
* Pregnancy
* Having a history of bariatric surgery
* Presence of contraindications to exercise testing

Inclusion Criteria for individuals with normal body mass index:

* Body mass index 18.5-24.9 kg/m2
* Volunteering for the study

Exclusion Criteria for individuals with normal body mass index:

* Body mass index > 25 kg/m2 or ≤18.5 kg/m2
* Having a known chronic or systemic disease
* Failure to cooperate with tests to be performed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with high and normal body mass index will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | 1st day
  It will be assessed by 6 minute pegboard and ring test.
Daily living activities | 1st day
  It will be evaluated with the Glittre activities of daily living test.

SECONDARY OUTCOMES:
Fatigue | 1st day
  Fatigue will be assessed with a Fatigue Severity scale. The scale consists of 9 questions.The total score ranges from 9 to 63. An average score of 4 and above indicates severe fatigue.
Pain | 1st day
  It will be evaluated with the Nordic Musculoskeletal Questionnaire. It consists of 27 items that assess the presence of musculoskeletal symptoms over a 12-month period, covering nine different parts of the body. There are also items on functional status and the presence of musculoskeletal symptoms in the last 7 days. The total number of painful areas is determined. Total number of painful areas varies from 0-9.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)